CLINICAL TRIAL: NCT05512403
Title: Evaluation of Diagnostic Performances of 18F-FDOPA PET KInetics as Biomarkers for the Improvement of Care of MRI Non-contrast Enhanced Gliomas
Brief Title: Evaluation of Diagnostic Performances of 18F-FDOPA PET KInetics
Acronym: KING
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, MD, PhD, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020PI126
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — fluorodopa F 18

STUDY DESIGN:
Intervention Model Description: Patients presenting with brain lesions that lack contrast enhancement on MRI, that are suspected to be LGGs and that are referred for biopsy or surgery within the following 6 months will be eligible for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Low Grade Glioma (LGG) without any MRI contrast enhancement (Experimental): Patients presenting with brain lesions that lack contrast enhancement on MRI, that are suspected to be LGGs and that are referred for biopsy or surgery within the following 6 months will be eligible for the study. The initial MRI should be performed a maximum of 3 weeks before patient inclusion and should at least include the conventional morphological sequences (T1, T1 sequences with injection of contrast product and T2 FLAIR).
  Patients will be selected in a neuro-oncological multidisciplinary consultation meeting.
  Interventions: Drug: PET/CT with 18F-DOPA

INTERVENTIONS:
Drug: PET/CT with 18F-DOPA — A 18F-FDOPA PET exam is then performed (acquisition of 30 minutes in List Mode format) according to the French guidelines for PET neuro-oncological indications (Verger et al. Med Nuc, 2020, (5)).
  Patient preparation and acquisition:
  * 4 hours of fasting
  * No carbidopa premedication
  * 2 MBq / kg of 18F-FDOPA
  * Dynamic acquisition in List Mode format for 30 min starting simultaneously with the patient's injection
  * Low dose scanner for attenuation correction

SUMMARY:
the investigators hypothesise that 18F-FDOPA PET kinetic parameters are good biomarkers to characterise suspected LGG brain lesions that exhibit no contrast on MRI, for identifying aggressive lesions. These parameters could constitute diagnostic biomarkers for this indication. This new diagnostic tool could enhance patient care in the short term in an evolving pathology affecting socially active subjects with a poor prognosis

DETAILED DESCRIPTION:
Diffuse low-grade gliomas (LGGs) without any contrast enhancement on MRI are rare (15% of gliomas, 700 cases/year in France), have a poor prognosis (median overall survival from 5 to 15 years) and affect young, socially active subjects (median age 40 years). Among these lesions, 30% present with high grade histopathological criteria or with poor prognostic molecular characteristics, according to the 2021 WHO Classification of Tumors of the Central Nervous System (lack of IDH [Isocitrate DeHydrogenase] mutation, CDKN2A/B deletion). These high-grade types of tumours progress within 6 months and their diagnosis and management represent a public health issue. Moreover, the care of LGG patients is currently not standardised.

Although treatment is based on surgery and the complete excision of the lesion, as far as this is possible, and/or first-line chemotherapy ±radiotherapy, the optimal time to begin treatment remains controversial.

Aggressive forms should be diagnosed as soon as possible to allow immediate surgery to improve survival, whilst strategies allowing the maintenance of an optimal quality of life, more often with functional surgery alone, are recommended for non-aggressive forms. The main hurdle to standardised patient management is the lack of amenable non-invasive biomarkers to identify aggressive LGG forms.

18F-FDOPA positron emission tomography (PET) is promising to diagnose initial gliomas with conventional Standardised-Uptake-Value (SUV) parameters. Our team recently demonstrated the potential of 18F-FDOPA PET kinetics to better characterise gliomas. Two parameters are determined from the 30-minute dynamic acquisition curve of the tumour: the time-to-peak SUV (TTP), and the SUV slope. In our previous studies, limited by their monocentric and retrospective nature, molecular characteristics were mainly predicted by TTP: long TTP for an IDH-mutation and short TTP for IDH-wildtype tumours. A prospective multicentric study is needed to confirm our preliminary results in a specific population of suspected LGGs without any contrast enhancement on MRI.

The investigator hypothesise that 18F-FDOPA PET kinetic parameters are biomarkers which lead to improved care because they characterise aggressive forms of gliomas exhibiting no contrast on MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old
* WHO general condition ≤2
* Identification of a unifocal brain tumour at the initial diagnosis with no contrast in the MRI and suspected to be a LGG, with biopsy/surgery envisaged within 6 months of the PET scan
* MRI performed a maximum of 3 weeks before inclusion and comprising the conventional morphological sequences (T1, T1 sequences with injection of contrast agent and T2 FLAIR).
* Subject affiliated to or beneficiary of a social security plan
* Subject having received complete information on the organisation of the research and having signed the informed consent form.

Exclusion Criteria:

* Multifocal brain lesions
* Contraindication to 18F-FDOPA PET
* Pregnant, parturient women or nursing mothers under Article L1121-5
* Women of childbearing age who do not have effective contraception under Article L1121-5
* Monitoring not possible
* Persons deprived of their liberty by a judicial or administrative decision under Article 1121-8, persons undergoing psychiatric treatment under Articles L. 3212-1 and L. 3213-1.
* Patients cannot simultaneously participate in an interventional research trial for the duration of the KING study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
To assess diagnostic performances of 18F-FDOPA PET (Positon Emission Tomography) Time-To-Peak in suspected LGGs without MRI -contrast enhancement for characterisation of aggressive lesions | 24 months
  the sensitivity, specificity, predictive positive value (PPV) and negative predictive value (NPV) of the 18F-FDOPA kinetic TTP parameter, to characterise aggressive lesions within suspected LGGs with no contrast enhancement on MRI at the initial diagnosis.

SECONDARY OUTCOMES:
To assess the diagnostic performances of 18F-FDOPA "slope", to characterise aggressive lesions | 24 months
  Sensitivity, specificity, Positive Predictive Value and Negative Predicitive Value of the 18F-FDOPA kinetic "slope" parameter
To assess the diagnostic performances of 18F-FDOPA SUV static conventional parameters and/or radiomics analyses associated with TTP kinetic parameter, to characterise aggressive lesions | 24 months
  Sensitivity, specificity, positive predictive and negative predictive values of the 18F-FDOPA conventional parameters and/or radiomics analysis and the kinetic parameter.
To assess, in patients suspected to have a non-contrast enhanced glioma at diagnosis the prevalence of aggressive forms within the suspected LGGs without any MRI contrast | 24 months
  Proportion of aggressive lesions expressed as an instantaneous prevalence and its 95% confidence interval of the total number of suspected LGGs without any contrast enhancement on MRI examined at initial diagnosis and referred for biopsy or surgery within the following 6 months.
  enhancement
To assess, in patients suspected to have a non-contrast enhanced glioma at diagnosis the clinical impact of the 18F-FDOPA PET (positon emission tomography) Time-To-Peak parameter | 24 months
  Number of patients who need to be diagnosed with 18F-FDOPA kinetic parameter TTP to identify an aggressive lesion within the suspected LGG population that do not exhibit any contrast enhancement on MRI at initial diagnosis and that undergo biopsy/surgery, defined as: 1/ [% of aggressive lesions detected with the 18F-FDOPA Time-To-Peak parameter].

CONTACTS AND LOCATIONS:
Overall Officials: Antoine VERGER, MD, PhD, Principal Investigator — CHRU Nancy; Aurélie KAS, MD, PhD, Principal Investigator — APHP salpêtrière PARIS; Eric GUEDJ, MD,PhD, Principal Investigator — APHM Marseille; Caroline BUND, MD, Principal Investigator — Institut de cancérologie Strasbourg Europe; Florence LEJEUNE, MD, PhD, Principal Investigator — Eugène MARQUIS Nantes; Anthelme FLAUS, MD, Principal Investigator — Hospices Civils de Lyon; Nicolas De LEIRIS, MD, Principal Investigator — University Hospital, Grenoble; Solène QUERELLOU, MD, Principal Investigator — CHRU de Brest; Laurent COLLOMBIER, MD, Principal Investigator — CHU de Nimes; Maria RIBEIRO, MD, PhD, Principal Investigator — CHU de Tours; Franck SEMAH, MD, PhD, Principal Investigator — CHU de Lille; Merwan GINET, MD, Principal Investigator — CHR Metz
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France